CLINICAL TRIAL: NCT03951233
Title: Genotyping K-RAS and EGFR in Greek Non-small-cell Lung Cancer Patients: Incidence, Significance and Treatment Implications
Brief Title: K-RAS and EGFR in Lung Cancer
Acronym: K-RAS_NSCLC
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: K-RAS_NSCLC
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin- fixed paraffin- embedded tissue blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- K-RAS and EGFR mutated
- Wild type

SUMMARY:
Retrospective analysis where patients with histologically confirmed Non-small cell lung cancer (NSCLC) were centrally evaluated for the presence of KRAS and EGFR mutations.

DETAILED DESCRIPTION:
A retrospective analysis, performed by the Hellenic Co-operative Oncology Group (HeCOG), in samples from patients with histologically confirmed NSCLC, who had been treated within HeCOG-affiliated centres from March 2000 through December 2012, were centrally evaluated for the presence of KRAS and EGFR mutations. All patients had available clinicopathological data at diagnosis. Formalin-fixed, paraffin-embedded tissue blocks were retrospectively retrieved from the HeCOG tumor repository. Cytologic material was prospectively submitted for genotyping in more recent years (2010-2012).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed NSCLC
* Signed and dated written informed consent
* Age 18 years
* Available cytological material

Exclusion Criteria: -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated within HeCOG-affiliated centres from March 2000 through December 2012.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2000-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | from the date of treatment start until verified disease progression, death from any cause or date of last contact whichever occurred first, up to 9 months
Overall survival | from the date of treatment start until verified disease progression, death from any cause or date of last contact whichever occurred first, up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Unit, Metropolitan Hospital, Neo Faliro, Athens, Greece

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Soda M, Choi YL, Enomoto M, Takada S, Yamashita Y, Ishikawa S, Fujiwara S, Watanabe H, Kurashina K, Hatanaka H, Bando M, Ohno S, Ishikawa Y, Aburatani H, Niki T, Sohara Y, Sugiyama Y, Mano H. Identification of the transforming EML4-ALK fusion gene in non-small-cell lung cancer. Nature. 2007 Aug 2;448(7153):561-6. doi: 10.1038/nature05945. Epub 2007 Jul 11. PMID 17625570
- [Background] Tan DS, Yom SS, Tsao MS, Pass HI, Kelly K, Peled N, Yung RC, Wistuba II, Yatabe Y, Unger M, Mack PC, Wynes MW, Mitsudomi T, Weder W, Yankelevitz D, Herbst RS, Gandara DR, Carbone DP, Bunn PA Jr, Mok TS, Hirsch FR. The International Association for the Study of Lung Cancer Consensus Statement on Optimizing Management of EGFR Mutation-Positive Non-Small Cell Lung Cancer: Status in 2016. J Thorac Oncol. 2016 Jul;11(7):946-63. doi: 10.1016/j.jtho.2016.05.008. Epub 2016 May 23. PMID 27229180
- [Background] Shepherd FA, Tsao MS. Unraveling the mystery of prognostic and predictive factors in epidermal growth factor receptor therapy. J Clin Oncol. 2006 Mar 1;24(7):1219-20; author reply 1220-1. doi: 10.1200/JCO.2005.04.4420. No abstract available. PMID 16505443
- [Background] Zhang Z, Wang T, Zhang J, Cai X, Pan C, Long Y, Chen J, Zhou C, Yin X. Prognostic value of epidermal growth factor receptor mutations in resected non-small cell lung cancer: a systematic review with meta-analysis. PLoS One. 2014 Aug 27;9(8):e106053. doi: 10.1371/journal.pone.0106053. eCollection 2014. PMID 25162713
- [Background] Pesek M, Benesova L, Belsanova B, Mukensnabl P, Bruha F, Minarik M. Dominance of EGFR and insignificant KRAS mutations in prediction of tyrosine-kinase therapy for NSCLC patients stratified by tumor subtype and smoking status. Anticancer Res. 2009 Jul;29(7):2767-73. PMID 19596959
- [Background] Satoh T, Nakafuku M, Kaziro Y. Function of Ras as a molecular switch in signal transduction. J Biol Chem. 1992 Dec 5;267(34):24149-52. No abstract available. PMID 1447166
- [Background] Wood K, Hensing T, Malik R, Salgia R. Prognostic and Predictive Value in KRAS in Non-Small-Cell Lung Cancer: A Review. JAMA Oncol. 2016 Jun 1;2(6):805-12. doi: 10.1001/jamaoncol.2016.0405. PMID 27100819
- [Background] Garassino MC, Marabese M, Rusconi P, Rulli E, Martelli O, Farina G, Scanni A, Broggini M. Different types of K-Ras mutations could affect drug sensitivity and tumour behaviour in non-small-cell lung cancer. Ann Oncol. 2011 Jan;22(1):235-237. doi: 10.1093/annonc/mdq680. No abstract available. PMID 21169473
- [Background] Ihle NT, Byers LA, Kim ES, Saintigny P, Lee JJ, Blumenschein GR, Tsao A, Liu S, Larsen JE, Wang J, Diao L, Coombes KR, Chen L, Zhang S, Abdelmelek MF, Tang X, Papadimitrakopoulou V, Minna JD, Lippman SM, Hong WK, Herbst RS, Wistuba II, Heymach JV, Powis G. Effect of KRAS oncogene substitutions on protein behavior: implications for signaling and clinical outcome. J Natl Cancer Inst. 2012 Feb 8;104(3):228-39. doi: 10.1093/jnci/djr523. Epub 2012 Jan 13. PMID 22247021
- [Background] Lee T, Lee B, Choi YL, Han J, Ahn MJ, Um SW. Non-small Cell Lung Cancer with Concomitant EGFR, KRAS, and ALK Mutation: Clinicopathologic Features of 12 Cases. J Pathol Transl Med. 2016 May;50(3):197-203. doi: 10.4132/jptm.2016.03.09. Epub 2016 Apr 18. PMID 27086595
- [Background] Lee B, Lee T, Lee SH, Choi YL, Han J. Clinicopathologic characteristics of EGFR, KRAS, and ALK alterations in 6,595 lung cancers. Oncotarget. 2016 Apr 26;7(17):23874-84. doi: 10.18632/oncotarget.8074. PMID 26992209
- [Background] Riely GJ, Kris MG, Rosenbaum D, Marks J, Li A, Chitale DA, Nafa K, Riedel ER, Hsu M, Pao W, Miller VA, Ladanyi M. Frequency and distinctive spectrum of KRAS mutations in never smokers with lung adenocarcinoma. Clin Cancer Res. 2008 Sep 15;14(18):5731-4. doi: 10.1158/1078-0432.CCR-08-0646. PMID 18794081
- [Background] Shepherd FA, Domerg C, Hainaut P, Janne PA, Pignon JP, Graziano S, Douillard JY, Brambilla E, Le Chevalier T, Seymour L, Bourredjem A, Le Teuff G, Pirker R, Filipits M, Rosell R, Kratzke R, Bandarchi B, Ma X, Capelletti M, Soria JC, Tsao MS. Pooled analysis of the prognostic and predictive effects of KRAS mutation status and KRAS mutation subtype in early-stage resected non-small-cell lung cancer in four trials of adjuvant chemotherapy. J Clin Oncol. 2013 Jun 10;31(17):2173-81. doi: 10.1200/JCO.2012.48.1390. Epub 2013 Apr 29. PMID 23630215
- [Background] Steuer CE, Behera M, Berry L, Kim S, Rossi M, Sica G, Owonikoko TK, Johnson BE, Kris MG, Bunn PA, Khuri FR, Garon EB, Ramalingam SS. Role of race in oncogenic driver prevalence and outcomes in lung adenocarcinoma: Results from the Lung Cancer Mutation Consortium. Cancer. 2016 Mar 1;122(5):766-72. doi: 10.1002/cncr.29812. Epub 2015 Dec 22. PMID 26695526
- [Background] Kotoula V, Charalambous E, Biesmans B, Malousi A, Vrettou E, Fountzilas G, Karkavelas G. Targeted KRAS mutation assessment on patient tumor histologic material in real time diagnostics. PLoS One. 2009 Nov 4;4(11):e7746. doi: 10.1371/journal.pone.0007746. PMID 19888477
- [Background] Altman DG, McShane LM, Sauerbrei W, Taube SE. Reporting Recommendations for Tumor Marker Prognostic Studies (REMARK): explanation and elaboration. PLoS Med. 2012;9(5):e1001216. doi: 10.1371/journal.pmed.1001216. Epub 2012 May 29. PMID 22675273
- [Background] Zhang YL, Yuan JQ, Wang KF, Fu XH, Han XR, Threapleton D, Yang ZY, Mao C, Tang JL. The prevalence of EGFR mutation in patients with non-small cell lung cancer: a systematic review and meta-analysis. Oncotarget. 2016 Nov 29;7(48):78985-78993. doi: 10.18632/oncotarget.12587. PMID 27738317
- [Background] Barlesi F, Mazieres J, Merlio JP, Debieuvre D, Mosser J, Lena H, Ouafik L, Besse B, Rouquette I, Westeel V, Escande F, Monnet I, Lemoine A, Veillon R, Blons H, Audigier-Valette C, Bringuier PP, Lamy R, Beau-Faller M, Pujol JL, Sabourin JC, Penault-Llorca F, Denis MG, Lantuejoul S, Morin F, Tran Q, Missy P, Langlais A, Milleron B, Cadranel J, Soria JC, Zalcman G; Biomarkers France contributors. Routine molecular profiling of patients with advanced non-small-cell lung cancer: results of a 1-year nationwide programme of the French Cooperative Thoracic Intergroup (IFCT). Lancet. 2016 Apr 2;387(10026):1415-1426. doi: 10.1016/S0140-6736(16)00004-0. Epub 2016 Jan 15. PMID 26777916
- [Background] Szumera-Cieckiewicz A, Olszewski WT, Tysarowski A, Kowalski DM, Glogowski M, Krzakowski M, Siedlecki JA, Wagrodzki M, Prochorec-Sobieszek M. EGFR mutation testing on cytological and histological samples in non-small cell lung cancer: a Polish, single institution study and systematic review of European incidence. Int J Clin Exp Pathol. 2013 Nov 15;6(12):2800-12. eCollection 2013. PMID 24294366
- [Background] Papadopoulou E, Tsoulos N, Tsirigoti A, Apessos A, Agiannitopoulos K, Metaxa-Mariatou V, Zarogoulidis K, Zarogoulidis P, Kasarakis D, Kakolyris S, Dahabreh J, Vlastos F, Zoublios C, Rapti A, Papageorgiou NG, Veldekis D, Gaga M, Aravantinos G, Karavasilis V, Karagiannidis N, Nasioulas G. Determination of EGFR and KRAS mutational status in Greek non-small-cell lung cancer patients. Oncol Lett. 2015 Oct;10(4):2176-2184. doi: 10.3892/ol.2015.3600. Epub 2015 Aug 12. PMID 26622815
- [Background] Mountzios G, Linardou H, S. A, editors. Epidemiology and incidence of EGFR mutation in Greek patients with advanced NSCLC. National Hellenic Oncology Meeting; 2016.
- [Background] Linardou H, Dahabreh IJ, Bafaloukos D, Kosmidis P, Murray S. Somatic EGFR mutations and efficacy of tyrosine kinase inhibitors in NSCLC. Nat Rev Clin Oncol. 2009 Jun;6(6):352-66. doi: 10.1038/nrclinonc.2009.62. PMID 19483740
- [Background] Murray S, Timotheadou E, Linardou H, Vrettou AV, Kostopoulos I, Skrickova J, Papakostantinou C, Christodoulou C, Pectasides D, Samantas E, Papakostas P, Skarlos DV, Kosmidis P, Fountzilas G. Mutations of the epidermal growth factor receptor tyrosine kinase domain and associations with clinicopathological features in non-small cell lung cancer patients. Lung Cancer. 2006 May;52(2):225-33. doi: 10.1016/j.lungcan.2005.12.015. Epub 2006 Mar 29. PMID 16567021
- [Background] Linardou H, Briasoulis E, Dahabreh IJ, Mountzios G, Papadimitriou C, Papadopoulos S, Bafaloukos D, Kosmidis P, Murray S. All about KRAS for clinical oncology practice: gene profile, clinical implications and laboratory recommendations for somatic mutational testing in colorectal cancer. Cancer Treat Rev. 2011 May;37(3):221-33. doi: 10.1016/j.ctrv.2010.07.008. Epub 2010 Sep 29. PMID 20817364
- [Background] Jung KJ, Jeon C, Jee SH. The effect of smoking on lung cancer: ethnic differences and the smoking paradox. Epidemiol Health. 2016 Dec 20;38:e2016060. doi: 10.4178/epih.e2016060. eCollection 2016. PMID 28092929
- [Background] Rulli E, Marabese M, Torri V, Farina G, Veronese S, Bettini A, Longo F, Moscetti L, Ganzinelli M, Lauricella C, Copreni E, Labianca R, Martelli O, Marsoni S, Broggini M, Garassino MC; TAILOR trialists. Value of KRAS as prognostic or predictive marker in NSCLC: results from the TAILOR trial. Ann Oncol. 2015 Oct;26(10):2079-84. doi: 10.1093/annonc/mdv318. Epub 2015 Jul 24. PMID 26209642
- [Background] Mascaux C, Iannino N, Martin B, Paesmans M, Berghmans T, Dusart M, Haller A, Lothaire P, Meert AP, Noel S, Lafitte JJ, Sculier JP. The role of RAS oncogene in survival of patients with lung cancer: a systematic review of the literature with meta-analysis. Br J Cancer. 2005 Jan 17;92(1):131-9. doi: 10.1038/sj.bjc.6602258. PMID 15597105
- [Background] Sun JM, Hwang DW, Ahn JS, Ahn MJ, Park K. Prognostic and predictive value of KRAS mutations in advanced non-small cell lung cancer. PLoS One. 2013 May 28;8(5):e64816. doi: 10.1371/journal.pone.0064816. Print 2013. PMID 23724098
- [Background] Linardou H, Dahabreh IJ, Kanaloupiti D, Siannis F, Bafaloukos D, Kosmidis P, Papadimitriou CA, Murray S. Assessment of somatic k-RAS mutations as a mechanism associated with resistance to EGFR-targeted agents: a systematic review and meta-analysis of studies in advanced non-small-cell lung cancer and metastatic colorectal cancer. Lancet Oncol. 2008 Oct;9(10):962-72. doi: 10.1016/S1470-2045(08)70206-7. Epub 2008 Sep 17. PMID 18804418
- [Background] Svaton M, Fiala O, Pesek M, Bortlicek Z, Minarik M, Benesova L, Topolcan O. The Prognostic Role of KRAS Mutation in Patients with Advanced NSCLC Treated with Second- or Third-line Chemotherapy. Anticancer Res. 2016 Mar;36(3):1077-82. PMID 26977001
- [Background] Bonanno L, Schiavon M, Nardo G, Bertorelle R, Bonaldi L, Galligioni A, Indraccolo S, Pasello G, Rea F, Favaretto A. Prognostic and predictive implications of EGFR mutations, EGFR copy number and KRAS mutations in advanced stage lung adenocarcinoma. Anticancer Res. 2010 Dec;30(12):5121-8. PMID 21187500
- [Background] Fan G, Zhang K, Ding J, Li J. Prognostic value of EGFR and KRAS in circulating tumor DNA in patients with advanced non-small cell lung cancer: a systematic review and meta-analysis. Oncotarget. 2017 May 16;8(20):33922-33932. doi: 10.18632/oncotarget.15412. PMID 28430611
- [Background] Shen H, Che K, Cong L, Dong W, Zhang T, Liu Q, Du J. Diagnostic and prognostic value of blood samples for KRAS mutation identification in lung cancer: a meta-analysis. Oncotarget. 2017 May 30;8(22):36812-36823. doi: 10.18632/oncotarget.15972. PMID 28415658
- [Background] Lohinai Z, Klikovits T, Moldvay J, Ostoros G, Raso E, Timar J, Fabian K, Kovalszky I, Kenessey I, Aigner C, Renyi-Vamos F, Klepetko W, Dome B, Hegedus B. KRAS-mutation incidence and prognostic value are metastatic site-specific in lung adenocarcinoma: poor prognosis in patients with KRAS mutation and bone metastasis. Sci Rep. 2017 Jan 4;7:39721. doi: 10.1038/srep39721. PMID 28051122
- [Background] Zhao N, Wilkerson MD, Shah U, Yin X, Wang A, Hayward MC, Roberts P, Lee CB, Parsons AM, Thorne LB, Haithcock BE, Grilley-Olson JE, Stinchcombe TE, Funkhouser WK, Wong KK, Sharpless NE, Hayes DN. Alterations of LKB1 and KRAS and risk of brain metastasis: comprehensive characterization by mutation analysis, copy number, and gene expression in non-small-cell lung carcinoma. Lung Cancer. 2014 Nov;86(2):255-61. doi: 10.1016/j.lungcan.2014.08.013. Epub 2014 Aug 30. PMID 25224251
- [Background] Mellema WW, Dingemans AM, Thunnissen E, Snijders PJ, Derks J, Heideman DA, Van Suylen R, Smit EF. KRAS mutations in advanced nonsquamous non-small-cell lung cancer patients treated with first-line platinum-based chemotherapy have no predictive value. J Thorac Oncol. 2013 Sep;8(9):1190-5. doi: 10.1097/JTO.0b013e318298764e. PMID 23787801
- [Background] Dong X, Zhao X, Hao Y, Wei Y, Yin Q, Du J. Response to first-line chemotherapy in patients with non-small-cell lung cancer according to epidermal growth factor receptor and K-RAS mutation status. Clin Lung Cancer. 2013 Nov;14(6):680-7. doi: 10.1016/j.cllc.2013.05.004. Epub 2013 Jul 31. PMID 23910066
- [Background] Marabese M, Ganzinelli M, Garassino MC, Shepherd FA, Piva S, Caiola E, Macerelli M, Bettini A, Lauricella C, Floriani I, Farina G, Longo F, Bonomi L, Fabbri MA, Veronese S, Marsoni S, Broggini M, Rulli E. KRAS mutations affect prognosis of non-small-cell lung cancer patients treated with first-line platinum containing chemotherapy. Oncotarget. 2015 Oct 20;6(32):34014-22. doi: 10.18632/oncotarget.5607. PMID 26416458
- [Background] Zhang Y, Fang W, Yan Y, Wang M, Kang S, Sheng J, Zhan J, Chen N, Hong S, Yang Y, Ma Y, He D, Qin T, Zhou T, Tang Y, He X, Liang W, Zhang L. The efficacy of first-line chemotherapy is associated with KRAS mutation status in patients with advanced non-small cell lung cancer: a meta-analysis. Med Oncol. 2015 Mar;32(3):61. doi: 10.1007/s12032-015-0489-y. Epub 2015 Feb 8. PMID 25663066
- [Background] Kim JH, Kim HS, Kim BJ. Prognostic value of KRAS mutation in advanced non-small-cell lung cancer treated with immune checkpoint inhibitors: A meta-analysis and review. Oncotarget. 2017 Jul 18;8(29):48248-48252. doi: 10.18632/oncotarget.17594. PMID 28525386
- [Background] Arrieta O, Cardona AF, Corrales L, Campos-Parra AD, Sanchez-Reyes R, Amieva-Rivera E, Rodriguez J, Vargas C, Carranza H, Otero J, Karachaliou N, Astudillo H, Rosell R; CLICaP. The impact of common and rare EGFR mutations in response to EGFR tyrosine kinase inhibitors and platinum-based chemotherapy in patients with non-small cell lung cancer. Lung Cancer. 2015 Feb;87(2):169-75. doi: 10.1016/j.lungcan.2014.12.009. Epub 2014 Dec 18. PMID 25558790
- [Result] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008